CLINICAL TRIAL: NCT01560559
Title: Peroral Endoscopic Myotomy for Primary Esophageal Achalasia
Acronym: TAMEO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011.696
Record Dates: First submitted 2012-03-06; First posted 2012-03-22 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2012-03

CONDITIONS: Primary Achalasia
Keywords: Primary esophageal achalasia; endoscopic myotomy; high resolution manometry
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Peroral endoscopic myotomy
  Interventions: Procedure: Peroral endoscopic myotomy

INTERVENTIONS:
Procedure: Peroral endoscopic myotomy — An endoscopy is performed under anesthesia with orotracheal intubation. After submucosal saline injection, an entry point in the submucosal space is created at 10 cm above the cardia. The endoscope will create a 12cm long tunnel in the caudal direction by submucosal dissection, stopping at 2cm below cardia. Then the muscular circular internal layer is sectioned on a 9cm length, starting 3 cm below the submucosal entry point. At the end the submucosal entry point is closed with metallic clips. A scanner is performed after the procedure so as to check the esophageal wall integrity. Alimentation is progressively introduced at day 1.
  This is a study of a procedure - peroral endoscopic myotomy (POEM). No new, unapproved device is used. All endoscopic tools are already approved for endoscopic submucosal dissection and associated complications (hemorrhage or perforation): dissection knifes, hot biopsy forceps, endoscopic metallic clips.

SUMMARY:
Recommended therapies for esophageal achalasia are endoscopic pneumatic dilation and Heller-Dor surgical myotomy. Endoscopic myotomy has been recently proposed in human patient in expert centers in Japan, US and Germany. In theory, endoscopic myotomy is as effective as surgical myotomy but less invasive and more effective with less complications than endoscopic pneumatic dilation. Up to now, published studies have confirmed these expectations, with 100% efficacy and no clinically significant complications. The present clinical trial with study the security and efficacy of peroral endoscopic myotomy in primary achalasia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged over 18 years old
2. Patients who have signed the informed consent form before any study related procedure
3. Primary achalasia of the cardia with Eckardt score > 3
4. Non sigmoid achalasia or S1 sigmoid type achalasia at barium meal Rx study
5. ASA score (American Society of Anaesthesiologists) 1 or 2
6. Patients affiliated to a social security health system

Exclusion Criteria:

1. Patients with age less than 18 years old
2. Patients without discernment with legal protection
3. Patients who will not be able to abide with study follow-up as judged by the investigator
4. Patients which cannot provide a written informed consent
5. Patient refusing to participate in the study, without informed consent
6. Pregnant or breastfeeding women, women in fertile age for procreation without efficient contraception, and/or positive serum βHCG test
7. Concomitant participation in other clinical trial
8. S2 sigmoid type primitive achalasia of the cardia
9. Pseudo-achalasia (esophageal carcinoma),
10. History of Barrett's esophagus with or without dysplasia, malignant tumors of the esophagus
11. History of esophageal strictures, systemic sclerosis
12. History of esophageal varices
13. History of endoscopic or surgical therapy of the esophageal achalasia
14. History of inferior endoscopic or surgical esophageal sphincter manipulation (sutures, polymers injection, adhesive bands)
15. History of surgical interventions of the esophagus or stomach (fundoplication, Heller-Dor myotomy, gastric resections, vagotomy with or without gastric drainage)
16. History of congenital of acquired coagulation anomalies: hemorrhagic diseases, hemostasis disturbances (TP < 60%, TCA > 40 seconds, platelets < 60000/mmc)
17. ASA score (American Society of Anaesthesiologists) 3, 4, 5 or 6
18. Cancer, liver, respiratory, renal or heart failure which put the patients in the ASA risk group 3,4,5 or 6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with clinically significant perforation | Day 1 after procedure
  Clinically significant perforation is defined as an ensemble of procedural, clinical, biological and imaging parameters:
  * perforation seen during procedure with placement of endoscopic metallic clips as closing method
  * acute severe persistent pain, fever over 38.5°C, subcutaneous emphysema, pneumomediastinum, penumoperitoneum
  * elevated white blood count with elevated neutrophils and elevated CRP, ascending values
  * subcutaneous emphysema, pneumomediastinum, penumoperitoneum seen at imaging studies (day 1 CT scan)

SECONDARY OUTCOMES:
percentage of patients with Eckardt score less than 3 | at 3rd and 12th month after procedure
  Eckardt score calculated at baseline and after procedure
significant variation of Eckardt score | at baseline and at 1st, 3rd, 6th and 12th month after the procedure
  Eckardt score calculated at baseline and after procedure
significant variation of GIQLI score | at baseline and at 1st, 3rd, 6th and 12th month after the procedure
  GIQLI score calculated at baseline and after procedure
significant variation of high resolution manometry parameters | at baseline and at 3rd month after the procedure
  high resolution manometry performed at baseline and at 3rd month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PONCHON, Pr, Principal Investigator — Hospices Civiles de Lyon
Locations (1):
- Clinique de Hépatogastroentérologie, Lyon, France